CLINICAL TRIAL: NCT03204396
Title: Smoking Cessation Facilitated by Glucagon-like Peptide-1 (GLP-1) Analogues - a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Smoking Cessation Facilitated by Glucagon-like Peptide-1 (GLP-1) Analogues
Acronym: SKIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-00286
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Glucagon-like Peptide-1; Smoking Cessation; Weight Change, Body; Craving
MeSH Terms: conditions — Smoking Cessation; Body Weight Changes | interventions — dulaglutide; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): Dulaglutide (Trulicity®) 1.5 mg in 0.5 ml, via pen s.c. once weekly for 12 weeks.
  Interventions: Drug: Dulaglutide
- Placebo group (Placebo Comparator): 0.5 ml normal saline (0.9% sodium chloride (NaCl)), injection s.c. via syringe once weekly for 12 weeks.
  Interventions: Drug: 0.5 ml normal saline (0.9% sodium chloride [0.9% NaCl])

INTERVENTIONS:
Drug: Dulaglutide — Application of Dulaglutide (Trulicity®) 1.5 mg s.c. once weekly for 12 weeks.
  Other Names: Trulicity
  Arms: Intervention group
Drug: 0.5 ml normal saline (0.9% sodium chloride [0.9% NaCl]) — Application of 0.5 ml normal saline (0.9% sodium chloride [0.9% NaCl]) once weekly for 12 weeks
  Arms: Placebo group

SUMMARY:
Cigarette smoking is the leading preventable cause of premature death worldwide. However smoking is a very difficult addiction to break whereby main reasons for not quitting or relapsing after cessation are the nicotine withdrawal syndrome and post-cessational weight gain. GLP-1 analogues are well known to stimulate insulin secretion and to reduce energy intake and therefore body weight. Recent findings from animal and human studies suggest a role of GLP-1 in the pathophysiology of addiction. The putative role of GLP-1 analogues in nicotine reward regulation combined with its weight reducing effects might be of major interest in view of novel pharmacotherapeutic options for smoking cessation.

* Substudy "fMRI": This substudy is to evaluate effects of Dulaglutide treatment on functional neuronal changes in smokers who want to quit smoking.
* Substudy "Energy": This substudy is to investigate the effect of Dulaglutide (Trulicity®) on REE and further parameters associated with energy metabolism (bodycomposition, haemodynamic parameters and catecholamine action) in a subset of patients recruited for the main trial.

DETAILED DESCRIPTION:
Cigarette smoking is the leading preventable cause of premature death worldwide. However smoking is a very difficult addiction to break and despite established smoking cessation programs quit rates are low, especially in the real-life setting. The main reasons for not quitting or relapsing after cessation are the nicotine withdrawal syndrome and post-cessational weight gain. GLP-1 analogues are well known to stimulate insulin secretion and to reduce energy intake and therefore body weight. Recent findings from animal and human studies suggest a role of GLP-1 in the pathophysiology of addiction. The putative role of GLP-1 analogues in nicotine reward regulation combined with its weight reducing effects might be of major interest in view of novel pharmacotherapeutic options for smoking cessation.

* Substudy "fMRI" (60 patients): Supposing that GLP-1 and analogues modulates nicotine induces reward system this substudy is to analyze if treatment with Dulaglutide (Trulicity®) attenuates craving and therefore functional brain activation. It is to evaluate effects of Dulaglutide treatment on functional neuronal changes in smokers who want to quit smoking.
* Substudy "Energy" (60 patients): The aim of the substudy "Energy" is to investigate the effect of Dulaglutide (Trulicity®) on REE and further parameters associated with energy metabolism (bodycomposition, haemodynamic parameters and catecholamine action) in a subset of patients recruited for the main trial.

ELIGIBILITY:
Inclusion Criteria for the main study:

* Age 18 to 75 years
* Daily smokers who are willing to quit and exhibit one of the following criteria: ≥10 cigarettes per day or
* At least moderate nicotine dependence defined by a Fagerstroem Score of ≥5 Points or
* Tobacco associated disease
* Treatment with varenicline (Champix®)

Additional Inclusion Criteria for the "substudy fMRI":

* Only patients aged 18-50 years are eligible

Additional Inclusion Criteria for the "substudy Energy":

* BMI of 18-30 kg/m2

Exclusion Criteria for the main study:

* Pregnancy (incl. wish to become pregnant within next 3 months) or breast feeding
* Pre-existing Treatment with GLP-1 agonists
* History of pancreatitis
* Severe renal insufficiency (estimated glomerular Filtration rate smaller than 30 ml/min/1.73 m2)
* Instable psychiatric conditions
* Anorexia nervosa

Additional Exclusion Criteria for the "substudy fMRI":

* Medical conditions that affect brain function (e.g. stroke, epilepsy, space occupying lesions, multiple sclerosis, Parkinson's disease, dementia, transient ischemic attack),
* Current use of medications that alter brain function
* Current illicit drug abuse including marijuana (alcohol ≤ 1 drink per day allowed)
* Claustrophobia, cardiac pacemaker, electronic device or ferromagnetic metal foreign bodies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Point prevalence abstinence rate at week 12 | 12 weeks
  Point prevalence abstinence rate at week 12 of dulaglutide treatment and Standard of care (SOC) versus SOC alone, confirmed with end-expiratory exhaled carbon monoxide measurements of 10 ppm or less

SECONDARY OUTCOMES:
Change in Body weight | 12 weeks
  Change in body weight in kg (and BMI [kg/m²]) relative to baseline at week 12 of dulaglutide treatment versus placebo.

OTHER OUTCOMES:
Point prevalence abstinence rate at week 24 and 52 | 52 weeks
  Point prevalence abstinence rate at weeks 24 and 52 of dulaglutide treatment and SOC versus SOC alone, confirmed with end-expiratory exhaled carbon monoxide measurements of 10 ppm or less
Prolonged abstinence rate at week 24 and 52 | 52 weeks
Smoking reduction at week 12, 24, and 52 | 52 weeks
Change of craving at week 4 and 12 relative to baseline | 12 weeks
Change of body weight in kg (and BMI [kg/m²]) at week 4, 8, 24, and 52 | 52 weeks
Change in haemoglobin A1c levels at week 12, 24, and 52 | 52 weeks
Craving measured by a Visual Analogue Scale (VAS) in the substudy "fMRI" | at week 12
  Behavioural endpoint of the substudy fMRI. The VAS rating scale includes seven steps from no craving to high craving.
Working memory performance investigated by the N-back task score in the substudy "fMRI" | at week 12
  Behavioural endpoint of the substudy fMRI. During the N-back task, all subjects see series of letters with an interstimulus interval of 2 s. Each stimulus is presented for 1 s. During a baseline (0-back) condition, subjects are required to press the button with the right hand when the letter "X" appears. During 1-back and 2-back conditions, participants are instructed to press the button if the currently presented letter is the same as that presented 1 (1-back condition) or 2 trials beforehand (2-back condition). The three conditions will be presented in ten alternating 30 s blocks (2 × 1-back, 3 × 2-back and 5 × 0-back) matched for the number of target letters per block (i.e., 2 or 3), in a pseudo-random order.
Blood oxygenated level dependent (BOLD) signal in fMRI in the substudy "fMRI" | at week 12
  Functional neuronal changes are assessed through the surrogate of blood oxygenated level dependent (BOLD) signal, an indirect measure of neural activity.
Change in structural plasticity of grey and white matter in fMRI in the substudy "fMRI" | at week 0 and at week 12
  Change in structural plasticity of grey and white matter in regions parts of the reward pathway (i.e. anterior cingulate cortex, insula, striatum) and in subcortical regions. One T1 sequence and one DTI sequence will be performed to investigate changes in grey and white matter.
Change of resting energy expenditure (REE) in the substudy "Energy" | at week 0 and at week 12
  Kcal per 24 hours. It is assessed by indirect calorimetry measuring volume of oxygen uptake (VO2) and expelled volume of carbon dioxide (VO2) in ml/min and calculated by the Weir Equation REE = [3.9 * (VO2) + 1.1 (VCO2)] * 1.44. The respiratory quotient (RQ) is calculated by dividing VCO2 by VO2.
Change in body composition in the substudy "Energy" | at week 0 and at week 12
  Body composition is assessed by bioelectrical impedance analysis. Measures are muscle and fat mass as a proportion (%) of total body weight.
Change in haemodynamic parameters in the substudy "Energy" | at week 0, 12, 24, 52
  Blood pressure (mmHg), heart rate (beats per minute), cardiac index (l/min/m2), and peripheral vascular resistance (Pa*[s/m3]) assessed by non-invasive thoracic bioimpedance (HOTMAN®)
Change in sympathetic activity in the substudy "Energy" | at week 0 and at week 12
  Plasma catecholamine (epinephrine and norepinephrine) and neuropeptide Y (NPY)* levels measured in pg/ml. NPY is a 36 aminoacid peptide well known to potentiate the action of catecholamine postsynaptically through the Y1 receptor and inhibit presynaptically the catecholamine secretion through the Y2 receptor

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Winzeler, Dr., Principal Investigator — University Hospital Basel, Endokrinology, diabetology, metabolism
Locations (1):
- Universitätsspital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beck J, Hasenbohler F, Werlen L, Lengsfeld S, Meienberg A, Bathelt C, Vogt D, Christ-Crain M, Burkard T, Winzeler B. Blood pressure changes during smoking cessation in a randomized, double-blind, placebo-controlled trial of dulaglutide treatment. Eur J Prev Cardiol. 2025 Oct 10;32(14):1394-1402. doi: 10.1093/eurjpc/zwaf055. PMID 40037282
- [Derived] Luthi H, Lengsfeld S, Burkard T, Meienberg A, Jeanloz N, Vukajlovic T, Bologna K, Steinmetz M, Bathelt C, Sailer CO, Laager M, Vogt DR, Hemkens LG, Speich B, Urwyler SA, Kuhne J, Baur F, Lutz LN, Erlanger TE, Christ-Crain M, Winzeler B. Effect of dulaglutide in promoting abstinence during smoking cessation: 12-month follow-up of a single-centre, randomised, double-blind, placebo-controlled, parallel group trial. EClinicalMedicine. 2024 Feb 9;68:102429. doi: 10.1016/j.eclinm.2024.102429. eCollection 2024 Feb. PMID 38371479
- [Derived] Baur F, Atila C, Lengsfeld S, Burkard T, Meienberg A, Bathelt C, Christ-Crain M, Winzeler B. Gender differences in weight gain during attempted and successful smoking cessation on dulaglutide treatment: a predefined secondary analysis of a randomised trial. BMJ Nutr Prev Health. 2023 Dec;6(2):301-309. doi: 10.1136/bmjnph-2023-000781. Epub 2023 Dec 19. PMID 38264360
- [Derived] Probst L, Monnerat S, Vogt DR, Lengsfeld S, Burkard T, Meienberg A, Bathelt C, Christ-Crain M, Winzeler B. Effects of dulaglutide on alcohol consumption during smoking cessation. JCI Insight. 2023 Nov 22;8(22):e170419. doi: 10.1172/jci.insight.170419. PMID 37991022
- [Derived] Lengsfeld S, Burkard T, Meienberg A, Jeanloz N, Coynel D, Vogt DR, Hemkens LG, Speich B, Zanchi D, Erlanger TE, Christ-Crain M, Winzeler B. Glucagon-like peptide-1 analogues: a new way to quit smoking? (SKIP)-a structured summary of a study protocol for a randomized controlled study. Trials. 2023 Apr 20;24(1):284. doi: 10.1186/s13063-023-07164-9. PMID 37081574
- [Derived] Lengsfeld S, Burkard T, Meienberg A, Jeanloz N, Vukajlovic T, Bologna K, Steinmetz M, Bathelt C, Sailer CO, Vogt DR, Hemkens LG, Speich B, Urwyler SA, Kuhne J, Baur F, Lutz LN, Erlanger TE, Christ-Crain M, Winzeler B. Effect of dulaglutide in promoting abstinence during smoking cessation: a single-centre, randomized, double-blind, placebo-controlled, parallel group trial. EClinicalMedicine. 2023 Feb 21;57:101865. doi: 10.1016/j.eclinm.2023.101865. eCollection 2023 Mar. PMID 36874396

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Substudy "SKIP-Energy" (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT03204396/Prot_SAP_000.pdf
  • Study Protocol: Appendix 4_SKIP Energy_V1_13_10_17 (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/96/NCT03204396/Prot_001.pdf
  • Study Protocol: Appendix 5_SKIP_Substudy fMRI (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/96/NCT03204396/Prot_002.pdf